CLINICAL TRIAL: NCT06773130
Title: An Exploratory Clinical Study of HRS-4642 Combined With Nimotuzumab in the Treatment of Recurrent or Metastatic Pancreatic Ductal Adenocarcinoma
Brief Title: HRS-4642 Combined With Nimotuzumab in the Treatment of Recurrent or Metastatic Pancreatic Ductal Adenocarcinoma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Dan Cao, Chief physician, West China Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PANC-2nd-IIT-HRS4642-NTZ
Record Dates: First submitted 2024-12-18; First posted 2025-01-14 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Pancreatic Ductal Adenocarcinoma (PDAC)
MeSH Terms: interventions — nimotuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HRS-4642+Nimotuzumab (Experimental): HRS-4642 in combination with Nimotuzumab, for recurrent or metastatic pancreatic ductal adenocarcinoma
  Interventions: Drug: HRS-4642; Drug: Nimotuzumab

INTERVENTIONS:
Drug: HRS-4642 — HRS-4642 will be administrated per dose level in which the patients are assigned.
Drug: Nimotuzumab — 400mg，ivgtt，d1，qw

SUMMARY:
To evaluate the safety and efficacy of HRS-4642 combined with Nimotuzumab in patients with recurrent or metastatic pancreatic ductal adenocarcinoma.

DETAILED DESCRIPTION:
This study is an open, single center, exploratory clinical trial aimed at evaluating the efficacy and safety of HRS-4642 combined with Nimotuzumab in the treatment of patients with recurrent or metastatic pancreatic ductal adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects aged 18-75 years (including 18 and 75 years).
2. Pancreatic ductal adenocarcinoma confirmed by pathology (histology) or cytology.
3. Patients with metastatic pancreatic ductal adenocarcinoma.
4. At the time of study enrollment, according to the solid tumor efficacy evaluation criteria (RECIST1.1), imaging diagnosis had at least one measurable lesion (lesion diameter ≥10 mm and lymph node diameter ≥15 mm according to CT or MRI evaluation).
5. Physical condition score ECOG score 0-2 points.
6. Expected survival ≥ 12 weeks.
7. Major organ function is normal.
8. The AE caused by previous anti-tumor therapy must be restored to the level of ≤ grade 1 (CTCAE v5.0) or the level specified in the inclusion criteria. If the investigator determines that NCI-CTCAE≤ grade 2 and there is no safety risk to the subject, the participant can be enrolled, such as receiving immune checkpoint inhibitor therapy. Subjects with type 1 diabetes and hypothyroidism that are stable after hormone replacement therapy.
9. Fertile female subjects must undergo a serum pregnancy test within 7 days before the first dose, and the result is negative; And must be non-lactating. Fertile female subjects and male subjects whose partners are women of reproductive age must agree to comply with the contraceptive requirement from the time of signing the informed consent until 30 days after the final administration of the trial drug (for subjects receiving HRS-4642);
10. The subjects voluntarily joined the study and signed the informed consent, with good compliance and follow-up.

Exclusion Criteria:

Patients will not be admitted to the study if they meet any of the following criteria:

1. The patient had previously used KRAS inhibitors or targeted EGFR therapy.
2. known allergy to the investigational drug or any of its components.
3. Systemic antitumor therapy (including unmarketed investigational drugs or therapies), such as chemotherapy, targeted therapy, and immunotherapy, has been received within 28 days prior to first administration, except for the following: oral fluorouracil and small-molecule targeted drugs within 14 days prior to first administration of investigational drugs or within 5 half-lives of drugs (whichever is longer). Chinese medicines with anti-tumor indications should be used within 14 days before the first use of the investigational drug; Surgical treatment (except diagnostic surgery) within 28 days prior to initial dosing; Patients who received local treatment such as radiotherapy, intervention or ablation within 14 days before the first dose.
4. Previous or concurrent suffering from other malignant tumors, Unless it is for basal cell carcinoma of the skin, superficial bladder cancer, squamous cell carcinoma of the skin, cervical carcinoma in situ, local prostate cancer, ductal carcinoma in situ of the breast after radical surgery, papillary carcinoma of the thyroid (allowing hormone therapy for non-metastatic prostate cancer or breast cancer) that has achieved complete remission at least 2 years prior to screening and does not require or is not expected to require other treatment during the study period;
5. accompanied by untreated or active central nervous system (CNS) tumor metastasis. Subjects with a history or current history of meningeal metastasis. Participants may be enrolled if their CNS metastases have been adequately localized (surgery or radiation) and do not require hormone therapy, and neurological recovery to baseline (except for lingering signs or symptoms associated with CNS treatment) is at least 2 weeks prior to initial treatment.
6. Patients with severe cardiovascular and cerebrovascular thromboembolism (e.g., myocardial infarction, unstable angina pectoris, stroke), NYHA grade 2 or above cardiac dysfunction, and clinically significant supratrioventricular or ventricular arrhythmias requiring clinical intervention in the 6 months prior to study entry.
7. Study the presence of digestive tract obstruction or signs and symptoms of digestive tract obstruction within 6 months prior to the start of treatment, but screening can be performed if surgical treatment has been performed, and the obstruction has been completely resolved.
8. Bleeding events of esophageal and gastric varices caused by portal hypertension occurred within 3 months before the first administration.
9. Had undergone a gastroscopy within 3 months prior to the first dose indicating severe (G3) varicose veins that were untreated or did not recover after treatment; There is current portal hypertension (including imaging evidence of splenomegaly) and the investigator determined that admission to the study would cause a greater risk of bleeding.
10. Advanced patients who are symptomatic, have spread to the internal organs, and are at risk of developing life-threatening complications in the short term (including patients with uncontrolled large exudates [chest, pericardium, abdominal cavity]); If effusion drainage is performed, patients who have been stable for at least 2 weeks after drainage can be enrolled in the group (local treatment within the serous cavity is allowed according to the diagnosis and treatment routine before signing the information).
11. Known or suspected pulmonary disease such as interstitial lung disease, non-infectious pneumonia, COPD, pulmonary embolism or other serious and uncontrolled medical disease, acute infection, recent history of major surgery (within 28 days or have not recovered from side effects).
12. Patients who had active tuberculosis infection within 1 year before enrollment or had a history of active tuberculosis infection more than 1 year before but had not received formal treatment.
13. Patients with congenital or acquired immune deficiency, such as human immunodeficiency virus (HIV) infection, active hepatitis B (HBV surface antigen [HBsAg] test positive during screening and HBV-DNA test value ≥10000 copies /ml [2000 IU/ml]), Active hepatitis C (positive for HCV antibody [HCV-AB] and HCV RNA during screening) or co-infection with hepatitis B and hepatitis C.
14. Acute or chronic pancreatitis with significant clinical significance; Patients at high risk for pancreatitis, such as those with serum amylase and/or lipase concentrations ≥3 ULN.
15. Use of live attenuated vaccine within 28 days prior to the initial study administration, or anticipated use of live attenuated vaccine during the study treatment.
16. Participated in a clinical trial of any drug or medical device within 4 weeks prior to initial dosing.
17. The presence of uncontrollable mental illness and other circumstances known to affect the completion of the study procedure, such as alcohol, drug or substance abuse, and criminal detention.
18. Other situations that the researchers believe should not be included.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-02-10 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
RP2D | Approximately 12 months
  RP2D will be determined on the basis of evaluation on safety and efficacy data in dose escalation stages.
ORR | Approximately 12 months
  ORR was evaluated by RECIST v1.1.

SECONDARY OUTCOMES:
DCR | 2 years
  Disease control rate (DCR) is assessed by investigators using RECIST 1.1 criteria.
DoR | 2 years
  Duration of response (DoR) is assessed by investigators using RECIST 1.1 criteria.
PFS | 2 years
  Progression-free survival (PFS) is assessed by investigators using RECIST 1.1 criteria.
OS | 2 years
  Overall survival (OS) is assessed by investigators using RECIST 1.1 criteria.
AEs | 2 years
  AEs are assessed by NCI-CTCAE v5.0

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital, Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Leng Q, Zhou J, Wang X, Zhang P, Xu H, Cao D. HRS-4642 combined with nimotuzumab in the treatment of recurrent or metastatic pancreatic ductal adenocarcinoma: study protocol of a single-arm, prospective phase Ib/II trial. Front Pharmacol. 2025 Jul 4;16:1562481. doi: 10.3389/fphar.2025.1562481. eCollection 2025. PMID 40689200